CLINICAL TRIAL: NCT03438435
Title: Fluorescence QRH-882260 Peptide Imaging in the Bile Duct
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: D. Kim Turgeon, MD (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Michael Saunders, MD, Clinical Professor of Medicine, University of Washington
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00130597
Record Dates: First submitted 2018-01-30; First posted 2018-02-19 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- QRH-882260 Heptapeptide (Experimental): Five mL of reconstituted (with sterile 0.9% NaCl) QRH-882260 Cy-5-labeled heptapeptide
  Interventions: Drug: QRH-882260 Heptapeptide

INTERVENTIONS:
Drug: QRH-882260 Heptapeptide — Imaging agent

SUMMARY:
Patients undergoing ERCP procedure with biliary stricture will have epithelial mucosa labeled with QRH-882260 fluorescence peptide that binds to EGFR. A custom mini-cholangioscope will be used to image the luminal surfaces of the biliary duct that are exposed to the fluorescence peptide. The images will be recorded and analyzed for relative fluorescence pattern and intensity and correlated to patient diagnosis and clinical outcomes.

DETAILED DESCRIPTION:
A Phase 1b study of the safety and efficacy of a topically-administered 7-amino acid peptide labeled with a near-infrared fluorophore Cy5 for detecting neoplastic areas of the bile duct is proposed. The study will test the safety and efficacy of administering this agent (QRH-882260 Heptapeptide) to human subjects undergoing clinically indicated ERCP for the evaluation of biliary disorders.

This is a pilot study of a single study group at a single center. The investigators intend to enroll 12 evaluable subjects. Expected enrollment is one subject every 1 month, so the study should take 12 to 24 months to complete. The expected duration of each subject's participation is 2 to 7 days.

Subjects will be recruited around their standard of care procedure. The endoscopists performing study procedures are all credentialed to do these procedures at the UWMC Digestive Health Center.

ERCP will proceed per UWMC standard of care. The endoscopists performing the procedure will evaluate the potential risk (if any) for the subject to continue with the study procedure. Five mL of the reconstituted QRH-882260 Heptapeptide (~100 μM) will be administered to the site of interest through a catheter in the standard endoscope. Five minutes after QRH-882260 Heptapeptide application, the unbound peptide will be washed off using the endogator irrigator and the residual liquid will be suctioned. Pictures with reflection-light and fluorescence will be taken with the SFE based molecular imaging mini-cholangioscope (MC) inserted via the instrument channel of the standard endoscope before the QRH-882260 Heptapeptide application, immediately after application and then again after the QRH-882260 Heptapeptide is rinsed.

The area of interest identified will be biopsied at the discretion of the endoscopist per clinical care. Any specimens taken will be for clinical care only and will be sent for routine histology per UWMC standard of care.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Male or female, aged 18 to 65
2. Scheduled for outpatient ERCP
3. Understands English and is interested in participating
4. Provides signed and dated informed consent form
5. Willing to comply with all study procedures and be available for the duration of the study

Exclusion Criteria:

1. Sleep apnea or respiratory problems
2. Pregnant or trying to conceive
3. Known allergy or negative reaction to components of the study product(s)
4. On active chemotherapy or radiation treatment
5. Anything that, in the opinion of the investigator, would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Treatment-related Adverse Events | 30 months
  Number of treatment-related Adverse Events when using fluorescent imaging with QRH during cholangioscopy

SECONDARY OUTCOMES:
Evaluation of imaging content based on the clinical diagnosis | 30 months
  Images taken during the procedure will be compared to the clinical diagnosis for the subject for correlation

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saunders, MD, Principal Investigator — Clinical Professor of Medicine
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No